CLINICAL TRIAL: NCT00638170
Title: The Efficacy of Cranberry Juice in the Prevention of Urinary Tract Infections in Children - Randomized, Placebo Controlled Multi-Center Study
Brief Title: Cranberry Juice in the Prevention of Urinary Tract Infections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Jarmo Salo/MD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 72/2001
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2008-01

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract Infections; Cranberry; Prevention
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Cranberry juice
  Interventions: Biological: Cranberry juice
- B (Placebo Comparator): Placebo juice
  Interventions: Biological: Placebo juice

INTERVENTIONS:
Biological: Cranberry juice — 5 ml/kg up to 300 ml, 1-2 doses daily for six months
  Arms: A
Biological: Placebo juice — 5 ml/kg up to 300 ml, 1-2 doses daily for six months
  Arms: B

SUMMARY:
The objective of the study is to determine whether recurrences of urinary tract infection in children can be prevented with cranberry juice.

DETAILED DESCRIPTION:
Five percent of children have at least one UTI episode and 30% of these episodes recur. Recurrences and the risk of renal damage are indications for long term antimicrobial prophylaxis, but emerging antimicrobial resistance underlines the need for alternatives. The bacteria causing urinary tract infection arise from the stools. Dietary changes can alter the balance of faecal bacteria. Vaccinium berries and products containing lactobacilli have been shown to act against the coliform bacteria that cause most urinary tract infections. In our previous study cranberry juice was effective in preventing symptomatic recurrences of urinary tract infections in women. The objective of our study is to determine whether recurrences of urinary tract infection in children can be prevented with cranberry juice.

ELIGIBILITY:
Inclusion Criteria:

* Urinary Tract Infection 0-2 months priorly

Exclusion Criteria:

* Antibiotic Prophylaxis

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 262 (Estimated)
Dates: Start 2001-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of the first recurrence | 12 months

SECONDARY OUTCOMES:
Total number of UTI episodes and use of antimicrobials | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matti Uhari, Professor, Study Director — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952